CLINICAL TRIAL: NCT01016600
Title: Phase I/II Trial of Azacitidine Plus Lenalidomide in the Treatment of Acute Myeloid Leukemia
Brief Title: Azacitidine and Lenalidomide for Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-1816 / 201101749
Record Dates: First submitted 2009-11-17; First posted 2009-11-19 (Estimated); Results first posted 2015-09-07 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-08

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Lenalidomide; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 (Experimental): Induction regimen (total 2 cycles)
  Lenalidomide 50 mg PO daily days 1-28
  Azacitidine 25 mg/m2 IV days 1-5
  Maintenance Regimen
  Lenalidomide 10 mg PO daily days 1-28
  Azacitidine 75 mg/m2 IV days 1-5
  Interventions: Drug: Lenalidomide; Drug: Azacitidine
- Cohort 2 (Experimental): Induction regimen (total 2 cycles)
  Lenalidomide 50 mg PO daily days 1-28
  Azacitidine 50 mg/m2 IV days 1-5
  Maintenance Regimen
  Lenalidomide 10 mg PO daily days 1-28
  Azacitidine 75 mg/m2 IV days 1-5
  Interventions: Drug: Lenalidomide; Drug: Azacitidine
- Cohort 3 (Experimental): Induction regimen (total 2 cycles)
  Lenalidomide 50 mg PO daily days 1-28
  Azacitidine 75 mg/m2 IV days 1-5
  Maintenance Regimen
  Lenalidomide 10 mg PO daily days 1-28
  Azacitidine 75 mg/m2 IV days 1-5
  Interventions: Drug: Lenalidomide; Drug: Azacitidine
- Phase II (Experimental): Induction regimen (total 2 cycles)
  Lenalidomide 50 mg PO daily days 1-28
  Azacitidine 75 mg/m2 (dose determined in Phase I) mg/m2 IV days 1-5
  Maintenance Regimen
  Lenalidomide 10 mg PO daily days 1-28
  Azacitidine 75 mg/m2 IV days 1-5
  Interventions: Drug: Lenalidomide; Drug: Azacitidine

INTERVENTIONS:
Drug: Lenalidomide
  Other Names: Revlimid
Drug: Azacitidine
  Other Names: Vidaza

SUMMARY:
Determine toxicity and remission rates of treatment with azacitidine and lenalidomide for patients with Acute Myeloid Leukemia

DETAILED DESCRIPTION:
Primary:

Phase 1:

To determine the toxicity and feasibility of combining lenalidomide and azacitidine in patients with relapsed/ refractory AML ≥ 18 years or untreated AML ≥60 years.

Phase 2:

To assess the complete remission (CRm plus CRi) rate after lenalidomide + azacitidine therapy in untreated AML ≥60 years.

Secondary:

1. To assess the response rate (RR), morphologic leukemia-free state, morphologic complete remission rate (CRm), cytogenetic CR (CRc) rate, CR with incomplete blood counts 14 rate, and partial remission 15 rate (PR).
2. To assess overall survival (OS) and event free survival (EFS).
3. To assess time to progression (TTP) in untreated AML ≥60 years.
4. To assess relapse free survival (RFS) and duration of CR for complete responders.
5. To determine the incidence and severity of other toxicities of lenalidomide in combination with azacitidine.
6. Assay the expression levels of cytokines/chemokines in the bone marrow plasma, expression of chemokine receptors/ligands on leukemic blasts important for the AML microenvironment and study the direct cytotoxic effects of lenalidomide, azacitidine and combination of both drugs on cryopreserved AML blast cells.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed AML age ≥ 60 years, de novo, secondary to prior therapy, or transformed from MDS, as defined by the International Working Group, except acute promyelocytic leukemia (AML M3) will be included for phase 1 and 2 study. Patients must not have abnormalities of inversion 16, t(16,16), del(16q), t(8,21) or t(15,17) as assessed by routine cytogenetics or FISH. Diagnosis of AML by WHO criteria (>20% blasts) is determined by CBC, bone marrow assessment, and immunophenotypic analysis performed within 2 weeks of study enrollment. No previous treatment for AML, however hydroxyurea, steroids, and leukopheresis are allowed.
* Relapsed AML age ≥18 years, except acute promyelocytic leukemia (AML M3), with CR < 1 years post 1st induction chemotherapy will be included in phase 1 study only.
* Primary refractory AML age ≥18 years, except acute promyelocytic leukemia (AML M3) post 1st induction chemotherapy will be included in phase 1 study only.
* Relapsed or refractory AML age ≥18 years, except acute promyelocytic leukemia (AML M3), post 1st salvage chemotherapy/ autologous stem transplantation/ allogeneic stem cell transplantation will be included in phase 1 study only.
* Understand and voluntarily sign an informed consent form.
* Able to adhere to the study visit schedule and other protocol requirements.
* ECOG performance status of ≤ 2 at study entry
* Life expectancy > 2 months
* WBC < 10,000 x 10^6/L (WBC counts may not be reduced by hydroxyurea or leukapheresis to achieve a WBC lower than 10,000 x 106 /L).
* Adequate renal and hepatic function as defined by:

  * Serum creatinine ≤ 1.5X institution ULN
  * Total bilirubin ≤ 2.0 mg/dL ( except Gilbert's syndrome or known hemolysis)
  * AST(SGOT) and ALT (SGPT) ≤ 2.5 x ULN
* All study participants must be registered into the mandatory Revlimid REMS® program, and be willing and able to comply with the requirements of Revlimid REMS®.
* Females of of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.
* Men must agree not to father a child and agree to use a latex condom during sexual contact with females of child bearing potential even if they have had a successful vasectomy. -Disease free of prior malignancies for ≥ 5 years with exception of AML, currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast.

Exclusion Criteria:

* Newly diagnosed AML age < 60 years.
* Newly diagnosed AML ≥ 60 years with favorable risk cytogenetic abnormalities as defined by SWOG criteria that include: inv(16)/t(16;16)/del(16q), t(15;17) with/without secondary aberrations, t(8;21) lacking del(9q) or complex karyotype 17. Prior to enrollment, FISH studies or routine cytogenetics must be completed to rule out these cytogenetic abnormalities.
* Known CNS leukemia
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Use of any other experimental drug or therapy within 30 days of enrollment.
* Known hypersensitivity to thalidomide and mannitol.
* The development of erythema multiforme if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Any prior use of lenalidomide
* Any prior use of azacytidine.
* Concurrent use of other anti-cancer agents or treatments (with the exception of steroids)
* Known positive for HIV or infectious hepatitis, type A, B or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-04; Primary Completion 2013-11 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Vij, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 31 participants were enrolled but only 30 participants started treatment and completed treatment.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Phase II
Started | 9 | 4 | 6 | 12
Completed | 8 | 4 | 6 | 12
Not Completed | 1 | 0 | 0 | 0
Not completed — Did not start treatment | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Phase II | Total
Number analyzed (Participants) | 9 | 4 | 6 | 12 | 31
Age, Continuous [Median (Full Range); unit: years] | 70 [64 to 74] | 67.5 [63 to 77] | 75.5 [65 to 81] | 72 [65 to 88] | 72 [63 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 3 | 4 | 14
  Male | 3 | 3 | 3 | 8 | 17
Region of Enrollment [Number; unit: participants]
  United States | 9 | 4 | 6 | 12 | 31

OUTCOME MEASURES:

1. Primary Outcome: Phase I Only - Maximum Tolerated Dose (MTD) as Measured by Dose-limiting Toxicities (DLTs)
Description: * The maximum tolerated dose (MTD) is defined as the dose level immediately below the dose level at which 2 patients of a cohort (of 2 to 6 patients) experience dose-limiting toxicity during the first cycle.
  * Hematologic DLT is as a persistent bone marrow aplasia with ≤ 10 % cellularity, which persists for > 60 days from the start of a chemotherapy cycle.
  * Non-hematologic DLT is defined as any Grade 3 or Grade 4 non-hematologic toxicity that occurs during the first cycle with the specific exceptions of nausea, vomiting, anorexia, weight loss, infections or electrolyte abnormalities attributable to any other cause. Grade 3 triglycerides will be considered a DLT only for patients who have Grade 3 in spite of appropriate lipid lowering drug therapy.
Time Frame: Completion of the phase I portion of study (approximately 1 year and 4 months)
Population: (1) participant in Cohort 1 did not start treatment. The Phase II cohort was not analyzed because this was a Phase I outcome only.
Measure: Number; unit: dose-limiting toxicities
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Phase II
Number analyzed (Participants) | 8 | 4 | 6 | 0
dose-limiting toxicities | 1 | 0 | 0 |

2. Primary Outcome: Phase I Only - Maximum Tolerated Dose (MTD)
Description: as for outcome 1
Time Frame: Completion of the phase I portion of study (approximately 1 year and 4 months)
Measure: Number; unit: mg/m^2
Groups:
- Phase I Cohort: Induction regimen (total 2 cycles)
  Lenalidomide 50 mg PO daily days 1-28
  Azacitidine 25 mg/m2 IV days 1-5
  Maintenance Regimen
  Lenalidomide 10 mg PO daily days 1-28
  Azacitidine 75 mg/m2 IV days 1-5
Arm/Group | Phase I Cohort
Number analyzed (Participants) | 18
mg/m^2 | 75

3. Secondary Outcome: Response Rate (CRm + CRc + CRi + PR)
Description: * Response rate (CRm + CRc + CRi + PR)
  * CRm = morphologic complete remission
  * CRc = cytogenetic complete remission
  * CRi = morphologic complete remission with incomplete blood count recovery
  * PR = partial remission
Time Frame: Median number of cycles completed [3 cycles (12 weeks) full range (1 (4 weeks)-17 (68 weeks))]
Population: (3) participants in Cohort 1, (1) participant in Cohort 2, and (3) participants in Phase II did not receive 28 days of lenalidomide and therefore are not evaluable for response. (1) participant in Cohort one had both CRm and CRc.
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Phase II
Number analyzed (Participants) | 5 | 3 | 6 | 9
participants
  CRm | 1 | 0 | 1 | 1
  CRc | 1 | 0 | 0 | 0
  CRi | 1 | 1 | 1 | 1
  PR | 2 | 0 | 2 | 5

4. Secondary Outcome: Morphologic Leukemia-free State
Description: Defined as < 5% blasts on the BM aspirate with spicules and a count of >200 nucleated cells and no blasts with Auer rods, and no persistent extramedullary disease.
Time Frame: Median number of cycles completed [3 cycles (12 weeks) full range (1 (4 weeks)-17 (68 weeks))]
Population: (3) participants in Cohort 1, (1) participant in Cohort 2, and (3) participants in Phase II did not receive 28 days of lenalidomide and therefore are not evaluable for response.
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Phase II
Number analyzed (Participants) | 5 | 3 | 6 | 9
participants | 2 | 1 | 2 | 2

5. Secondary Outcome: Morphologic Complete Remission Rate (CRm)
Description: Defined as morphologic leukemia-free state, including <5% blasts in BM aspirate with marrow spicules and a count of > 200 nucleated cells and no blasts with Auer rods, no persistent extramedullary disease, ANC > 1000/uL, platelet count > 100,000/uL. Patient must be independent of transfusions for a minimum of 1 week before each marrow assessment. There is no duration requirement for this designation.
Time Frame: Completion of treatment (median follow-up was 8 weeks) (range 4-68 weeks)
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Phase II
Number analyzed (Participants) | 5 | 3 | 6 | 9
participants | 1 | 0 | 1 | 1

6. Secondary Outcome: Cytogenetic CR (CRc) Rate
Description: Only patients with an identified cytogenetic abnormality may receive this designation. Defines as a morphologic complete remission plus reversion to a normal karyotype (no clonal abnormalities detected in a minimum of 20 mitotic cells).
Time Frame: Completion of treatment (median follow-up was 8 weeks) (range 4-68 weeks)
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Phase II
Number analyzed (Participants) | 5 | 3 | 6 | 9
participants | 1 | 0 | 0 | 0

7. Secondary Outcome: CR With Incomplete Blood Counts Rate
Description: Defined as CR with the exception of neutropenia <1000/uL or thrombocytopenia <100,000/ul.
Time Frame: Completion of treatment (median follow-up was 8 weeks) (range 4-68 weeks)
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Phase II
Number analyzed (Participants) | 5 | 3 | 6 | 9
participants | 1 | 1 | 1 | 1

8. Secondary Outcome: Partial Remission Rate (PR)
Description: Requires that the criteria for complete remission be met with the following exceptions: decrease of >50% in the percentage of blasts to 5-25% in the BM aspirate. A value of < 5% blasts in BM with Auer rods is also considered a partial remission.
Time Frame: Completion of treatment (median follow-up was 8 weeks) (range 4-68 weeks)
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Phase II
Number analyzed (Participants) | 5 | 3 | 6 | 9
participants | 2 | 0 | 2 | 5

9. Secondary Outcome: Overall Survival
Description: Defined as the date of first dose of study drug to the date of death from any cause.
Time Frame: Until death - median follow-up 4.6 months (full range (0.3-31.4 months))
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Phase II
Number analyzed (Participants) | 8 | 4 | 6 | 12
months | 4.2 [0.7 to 31.4] | 4.5 [0.7 to 10.6] | 8.9 [1.8 to 14.8] | 4.3 [0.8 to 31.0]

10. Secondary Outcome: Event Free Survival
Description: Defined as the interval from the date of first dose of study drug to date of treatment failure, recurrence, or death due to any cause.
Time Frame: Until death - median follow-up 4.6 months (full range (0.3-31.4 months))
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Phase II
Number analyzed (Participants) | 8 | 4 | 6 | 12
months | 3.8 [0.3 to 19.7] | 3.4 [0.6 to 6.4] | 7.8 [1.8 to 14.8] | 2.9 [0.8 to 25.6]

11. Secondary Outcome: Time to Progression (TTP)
Description: Defined as the interval from the date of the first dose of study drug to the date of progressive disease.
Time Frame: Until progressive disease - median follow-up 4.6 months (full range (0.3-31.4 months))
Population: (2) cohort 1 participants were not evaluable for this outcome measure because (1) was removed for DLT & (1) withdrew from study. (2) phase II participants were not evaluable because both were removed from study in the first cycle for adverse events.
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Phase II
Number analyzed (Participants) | 6 | 4 | 6 | 10
months | 5.7 [0.3 to 19.7] | 3.4 [0.6 to 6.4] | 7.8 [1.8 to 14.8] | 3.7 [0.9 to 25.6]

12. Secondary Outcome: Relapse Free Survival (RFS)
Description: This is determined only for patients achieving a complete remission. Defined as the interval from the date of first documentation of a leukemia free state to date of recurrence or death due to any cause.
Time Frame: Until death - median follow-up 4.6 months (full range (0.3-31.4 months))
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Phase II
Number analyzed (Participants) | 2 | 1 | 2 | 2
months | 12.0 [6.2 to 17.7] | 1.4 [1.4 to 1.4] | 4.9 [3.2 to 6.7] | 12.2 [1.1 to 23.2]

13. Secondary Outcome: Duration of CR for Complete Responders
Time Frame: Completion of treatment (median follow-up was 8 weeks) (range 4-68 weeks)
Population: (6) participants in Cohort 1, (3) participants in Cohort 2, (4) participants in Cohort 3, and (10) participants in Phase II did not have a complete response and are not evaluable for this outcome.
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Phase II
Number analyzed (Participants) | 2 | 1 | 2 | 2
months | 10.9 [6.2 to 15.6] | 1.4 [1.4 to 1.4] | 4.95 [3.2 to 6.7] | 12.15 [1.1 to 23.2]

14. Secondary Outcome: Toxicity Profile (Grade 3/4 Toxicities)
Description: AML ≥18 years or untreated AML ≥60 years
Time Frame: 30 days after completion of treatment (median follow-up was 12 weeks (range 8-72 weeks))
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Phase II
Number analyzed (Participants) | 8 | 4 | 6 | 12
participants
  Anemia | 3 | 0 | 0 | 4
  Febrile neutropenia | 4 | 1 | 3 | 8
  Otitis mastoditis - worsening | 1 | 0 | 0 | 0
  Diarrhea | 1 | 0 | 2 | 0
  Nausea | 1 | 0 | 0 | 1
  Vomiting | 2 | 0 | 0 | 2
  Dental carries | 1 | 0 | 0 | 0
  Fatigue | 1 | 0 | 4 | 4
  Sepsis | 1 | 0 | 2 | 1
  Bronchial infection | 1 | 0 | 0 | 0
  Bacteremia | 2 | 0 | 1 | 0
  Lung infection | 3 | 0 | 2 | 9
  Skin infection | 1 | 2 | 2 | 2
  Activated partial thromboplastin time prolonged | 1 | 0 | 0 | 0
  Blood bilirubin increased | 2 | 0 | 2 | 3
  Creatinine increased | 1 | 0 | 1 | 0
  Neutrophil count decreased | 7 | 0 | 2 | 2
  Platelet count decreased | 4 | 2 | 3 | 6
  White blood cell count decreased | 7 | 1 | 4 | 10
  Lymphocyte count decreased | 5 | 1 | 1 | 2
  Dehydration | 2 | 0 | 0 | 3
  Hypernatremia | 1 | 0 | 0 | 0
  Hypocalcemia | 1 | 0 | 1 | 0
  Hypophosphatemia | 4 | 0 | 3 | 6
  Back pain | 1 | 0 | 0 | 0
  Generalized muscle weakness | 2 | 0 | 1 | 2
  Pain in extremity | 1 | 0 | 0 | 1
  Leukemia vasculitis left calf | 1 | 0 | 0 | 0
  Acute kidney injury | 1 | 0 | 1 | 0
  Dyspnea | 3 | 2 | 1 | 2
  Epistaxis | 1 | 0 | 0 | 0
  Productive cough | 1 | 0 | 1 | 0
  Pulmonary edema | 1 | 0 | 0 | 0
  Rash maculo-papular | 1 | 0 | 1 | 1
  Skin ulceration | 1 | 0 | 0 | 0
  Hypotension | 3 | 0 | 1 | 1
  Constipation | 0 | 1 | 0 | 0
  Edema limbs | 0 | 1 | 0 | 1
  Catheter related infection | 0 | 1 | 1 | 1
  Alanine aminotransferase increased | 0 | 1 | 0 | 1
  INR increased | 0 | 1 | 0 | 0
  Hyperglycemia | 0 | 1 | 0 | 5
  Hematuria | 0 | 1 | 0 | 1
  Cough | 0 | 1 | 0 | 0
  Wheezing | 0 | 1 | 0 | 0
  Cardiac arrest | 0 | 0 | 1 | 0
  Perianal hemorrhage | 0 | 0 | 1 | 0
  Cyst infection | 0 | 0 | 1 | 0
  Incarcerated hernia | 0 | 0 | 1 | 0
  Hypoalbuminemia | 0 | 0 | 1 | 1
  Hypokalemia | 0 | 0 | 2 | 3
  Respiratory failure | 0 | 0 | 1 | 1
  Pruritus | 0 | 0 | 1 | 0
  Hypertension | 0 | 0 | 1 | 0
  Atrial fibrillation | 0 | 0 | 0 | 1
  Chest pain cardiac | 0 | 0 | 0 | 1
  Left ventricular systolic dysfunction | 0 | 0 | 0 | 1
  Supraventricular tachycardia | 0 | 0 | 0 | 1
  Dysphagia | 0 | 0 | 0 | 1
  Esophagitis | 0 | 0 | 0 | 1
  Lower gastrointestinal hemorrhage | 0 | 0 | 0 | 1
  Pain | 0 | 0 | 0 | 1
  Otitis media | 0 | 0 | 0 | 1
  Scrotal infection | 0 | 0 | 0 | 1
  Upper respiratory infection | 0 | 0 | 0 | 1
  Urinary tract infection | 0 | 0 | 0 | 1
  Wound infection | 0 | 0 | 0 | 1
  Fall | 0 | 0 | 0 | 1
  Fracture | 0 | 0 | 0 | 1
  Weight loss | 0 | 0 | 0 | 1
  Anorexia | 0 | 0 | 0 | 1
  Hyponatremia | 0 | 0 | 0 | 3
  Neck pain | 0 | 0 | 0 | 1
  Polyarthropathy | 0 | 0 | 0 | 1
  Syncope | 0 | 0 | 0 | 2
  Pleuritic pain | 0 | 0 | 0 | 2

15. Primary Outcome: Phase II Only - Complete Remission Rate (CRm + CRi) in Participants With Untreated AML ≥60 Years of Age
Description: * Morphologic complete remission (CRm): Defined as morphologic leukemia-free state, including <5% blasts in BM aspirate with marrow spicules and a count of > 200 nucleated cells and no blasts with Auer rods, no persistent extramedullary disease, ANC > 1000/uL, platelet count > 100,000/uL. Patient must be independent of transfusions for a minimum of 1 week before each marrow assessment.
  * Morphologic complete remission with incomplete blood count recovery (CRi): Defined as CR with the exception of neutropenia <1000/uL or thrombocytopenia <100,000/ul.
Time Frame: Completion of treatment (median follow-up was 8 weeks) (range 4-68 weeks)
Population: Participants in Cohort 1, 2, and 3 were not analyzed for this outcome as it is a Phase II outcome measure only. (3) participants in Phase II cohort were not evaluable for response because they did not complete cycle 1.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Phase II
Number analyzed (Participants) | 0 | 0 | 0 | 9
percentage of participants |  |  |  | 22

ADVERSE EVENTS:
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Phase II
Serious Adverse Events (participants affected / at risk) | 8/8 | 2/4 | 6/6 | 12/12
Other Adverse Events (participants affected / at risk) | 8/8 | 4/4 | 6/6 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=8) | Cohort 2 (N=4) | Cohort 3 (N=6) | Phase II (N=12)
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Bacteremia blood (Infections and infestations) | 2 | 0 | 1 | 0
Bleeding (General disorders) | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Catheter related infection (Infections and infestations) | 0 | 0 | 1 | 1
Confusion (Nervous system disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Cyst infection (Infections and infestations) | 0 | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Edema (General disorders) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1 | 0
Febrile neutropenia (Infections and infestations) | 3 | 0 | 1 | 3
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Hemorrhoidal hemorrage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hernia (General disorders) | 0 | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 3 | 0 | 1 | 0
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Itching (General disorders) | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 9
Otitis media (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Post operative hemorrhage (bone marrow biopsy site) (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Progressive disease (General disorders) | 2 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Scrotal infection (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Skin infection (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Thrombocytopenia (Investigations) | 1 | 0 | 0 | 0
Thromboembolic event DVT (Vascular disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=8) | Cohort 2 (N=4) | Cohort 3 (N=6) | Phase II (N=12)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 5
Activated partial thromboplastin time prolonged (Investigations) | 3 | 0 | 1 | 3
Acute gout attack (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 2 | 2
Acute systolic CHF/MV regurgitation (Cardiac disorders) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 5 | 3 | 3 | 9
Alkaline phosphatase increased (Investigations) | 4 | 1 | 3 | 4
Anemia (Blood and lymphatic system disorders) | 2 | 0 | 2 | 4
Anorexia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 5
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 4 | 1 | 1 | 6
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 5
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 3
Blood bilirubin increased (Investigations) | 4 | 0 | 4 | 8
Blurred vision (Eye disorders) | 0 | 0 | 0 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Bronchial infection (Infections and infestations) | 1 | 0 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 4
Cardiac troponin I increased (Investigations) | 0 | 0 | 0 | 1
Catheter related infection (Infections and infestations) | 0 | 1 | 0 | 0
Chest pain - cardiac (Cardiac disorders) | 0 | 0 | 0 | 1
Chills (General disorders) | 3 | 1 | 2 | 7
Clostridium difficile (Infections and infestations) | 0 | 0 | 0 | 1
Confusion (Psychiatric disorders) | 2 | 0 | 2 | 2
Constipation (Gastrointestinal disorders) | 3 | 1 | 1 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 6
Creatinine increased (Investigations) | 4 | 1 | 1 | 4
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 4 | 0 | 0 | 4
Delerium (Nervous system disorders) | 0 | 0 | 0 | 1
Dental carries (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 4 | 1 | 4 | 7
Dizziness (Nervous system disorders) | 2 | 3 | 0 | 3
Double vision (Eye disorders) | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 1 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 4 | 8
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Edema face (General disorders) | 0 | 0 | 0 | 1
Edema limbs (General disorders) | 6 | 0 | 3 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 3
Erythemia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Esophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Eye abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 1 | 0
Facial muscle weakness (Nervous system disorders) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2
Fatigue (General disorders) | 6 | 4 | 4 | 9
Febrile neutropenia (Infections and infestations) | 1 | 1 | 2 | 5
Fever (General disorders) | 3 | 0 | 0 | 1
Flashing lights (Eye disorders) | 0 | 0 | 0 | 1
Flu Like Symptoms (General disorders) | 0 | 0 | 0 | 1
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5 | 1 | 3 | 6
Gram positive cocci (Infections and infestations) | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 1 | 0 | 0 | 4
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 2
Hematoma (Vascular disorders) | 0 | 0 | 1 | 1
Hematuria (Renal and urinary disorders) | 1 | 1 | 1 | 6
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hot flashes (Vascular disorders) | 0 | 0 | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 1 | 1 | 4
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 4
Hypertension (Vascular disorders) | 1 | 0 | 1 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 | 2 | 2 | 11
Hypocalcemia (Metabolism and nutrition disorders) | 6 | 3 | 5 | 11
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 7
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 3 | 2 | 4 | 7
Hypophosphatemia (Metabolism and nutrition disorders) | 5 | 1 | 3 | 7
Hypotension (Vascular disorders) | 0 | 0 | 1 | 2
Hypothermia (General disorders) | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 2 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 6
INR increased (Investigations) | 2 | 1 | 1 | 8
Incarcerated hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Infusion related reaction (General disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 2
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0
Leukemia vasculitis left calf (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lip infection (Infections and infestations) | 1 | 0 | 0 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 5 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 5 | 1 | 4 | 9
Lymphocyte count increased (Investigations) | 0 | 0 | 0 | 1
Lytic lesion in right parietal bone (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 2
Mucositis - oral (Gastrointestinal disorders) | 2 | 1 | 2 | 8
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 3 | 5 | 8
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 7 | 0 | 2 | 2
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 2
Oral hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oral thrush (Infections and infestations) | 1 | 0 | 1 | 4
Otitis mastoiditis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 3 | 1 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Perianal hemorrhage (General disorders) | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1
Perirectal abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 3 | 2 | 3 | 7
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 4
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Polyarthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3 | 4
Proteinuria (Renal and urinary disorders) | 1 | 0 | 1 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 3 | 4
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 1 | 2 | 7
Rash-petechial (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rectal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Renal tubular acidosis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Scrotal infection (Infections and infestations) | 0 | 1 | 0 | 0
Scrotal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 2
Sepsis (Infections and infestations) | 1 | 0 | 1 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 1 | 4
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 3 | 3 | 2 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 3
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Splenomegaly (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Staphylococcus epidermis-blood (Infections and infestations) | 0 | 0 | 0 | 1
Stroke (Nervous system disorders) | 0 | 0 | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Systolic murmur (Cardiac disorders) | 0 | 0 | 1 | 0
Thromboembolic event (Vascular disorders) | 0 | 1 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 2
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 0 | 4
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 2
VRE stool (Infections and infestations) | 0 | 0 | 0 | 2
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Visual disturbance/double vision (Eye disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 2 | 4 | 7
Vulval infection (Infections and infestations) | 0 | 0 | 1 | 0
Weight gain (Investigations) | 0 | 0 | 0 | 1
Weight loss (Investigations) | 0 | 0 | 1 | 5
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
White blood cell decreased (Investigations) | 7 | 1 | 5 | 10
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes